CLINICAL TRIAL: NCT05528718
Title: Sustained Mood Improvement With Laughing Gas Exposure: A Randomized Controlled Pilot Trial - Sub-Study Protocol to Include Neuroimaging
Brief Title: SMILE Trial - Imaging Sub-Study
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-139
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Endothelium-Dependent Relaxing Factors; Inhalation; Midazolam; Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Participants assigned to this intervention arm in the main study will have been administered nitrous oxide at an inspiratory concentration of 50% with concurrent intravenous saline (100mL) for one hour.
  Interventions: Drug: Nitrous oxide gas for inhalation
- Placebo group: Participants assigned to this intervention arm in the main study will have been administered 50% oxygen with intravenous midazolam (0.02mg/kg in 100mL) for one hour.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Nitrous oxide gas for inhalation — This sub-study does not have an intervention and based on the main study the participants who have received N2O will be compared with the midazolam placebo group.
  Other Names: Nitrous oxide at an inspiratory concentration of 50% with concurrent intravenous saline (100mL)
  Groups: Experimental group
Drug: Midazolam injection — This sub-study does not have an intervention and based on the main study the participants who have received N2O will be compared with the midazolam placebo group.
  Other Names: 50% oxygen with intravenous midazolam (0.02mg/kg in 100mL)
  Groups: Placebo group

SUMMARY:
This is a pilot sub-study of an ongoing trial comparing N2O to midazolam in MDD and will examine neuroimaging correlates of treatment response.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) scans of MDD-affected brains have revealed changes in structural and functional connectivity compared to healthy subjects. This pilot sub-study examines structural and functional connectivity associated with MDD-affected patient participants' responsiveness to N2O compared to the midazolam placebo, which induces similar sedative effects. The investigators intend to address the changes in brain functional activity and connectivity between baseline and after a four-week intervention course involving weekly nitrous oxide inhalations measured by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for main nitrous oxide (SMILE) study

Exclusion Criteria:

* Contraindication for undergoing MRI scans (e.g., hip circumference < 180 cm or metal in the body)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient participants were diagnosed as suffering from major depressive disorder (MDD) that meets the criteria of the Diagnosis and Statistical Manual for Mental Disorders (DSM-5), will be eligible to participate in this data collection study. Participants who have agreed to receive N2O treatments as part of the Interventional Psychiatry Clinical Program at St. Michael's Hospital will be approached and recruited.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Brain functional activity and connectivity | 4 weeks from the baseline visit
  Changes in brain functional activity and connectivity between baseline and after 4 weeks of receiving the intervention, measured by MR imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Bhat, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No